CLINICAL TRIAL: NCT07318298
Title: Effect of Injectable Hyaluronic Acid (HYADENT BG (HA)) on Bone Healing in Extraction Sockets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 35/175/2024; 644/2024 (Other Grant/Funding Number: Jordan University of Science and Technology)
Record Dates: First submitted 2025-08-25; First posted 2026-01-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: The Application of Hyaluronic Acid on Teeth Bone Healing. Hyaluronic Acid Which is Widely Used in Medicine for Joint, Eye Care, Wound Healing
Keywords: hyauronic acid, wisdom teeth extraction, bone healing

STUDY DESIGN:
Intervention Model Description: application of Hyaluronic acid
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo extraction side (Placebo Comparator): Surgical extraction of wisdom tooth with placebo administration inside the extraction site using collagen sponge
  Interventions: Procedure: Surgical extraction of wisdom teeth; Procedure: bone biobsy
- experimental extraction side (Experimental): Surgical extraction of wisdom tooth with placebo administration inside the extraction site using hyaluronic acid gel
  Interventions: Procedure: Surgical extraction of wisdom teeth; Procedure: bone biobsy

INTERVENTIONS:
Procedure: Surgical extraction of wisdom teeth — A standardized surgical procedure was performed by a single experienced surgeon (ZA). Under strict aseptic conditions, an inferior alveolar nerve block with buccal infiltration, was given using lidocaine HCl 2% with epinephrine 1:100,000 (Cook-Waite, Rochester, NY). A mucoperiosteal envelope flap was utilized for all surgeries. Bone removal and tooth sectioning were performed as deemed necessary using a low-speed handpiece under copious saline irrigation. After tooth removal, HA gel (Hyadent) was placed inside the extraction socket and covered with collagen sponge in the test sockets, while only coverage with collagen sponge was placed in the control sockets. Subsequently, flap closure was achieved using 3-0 silk sutures
Procedure: bone biobsy — After 6 weeks, core biopsies are taken from both sides. Under local anesthesia, the core biopsies sre taken without reflection of a flap, using a graded trephine bur (MCT, Korea) of 3 mm diameter (which is not invasive or having any complication) for later histological evaluation. Specimens harvested from each patient are fixed in 10% formalin, then decalcified using 10% hydrochloric acid. After processing, 5 micrometer sections are prepared and stained with hematoxylin and eosin stain (H&E).
  Digital images are acquired from each section at a magnification of × 40. ImageJ 1.52a software (National Institute of Health, Bethesda, Maryland, USA) is used to calculate the percentage of woven bone area within selected regions of interest (ROI) in each image, utilizing the color thresholding feature. To ensure that measurements are valid, 3 measurements are made for each of the hard tissue and soft tissue components, and for the total area of the ROI in pixels.

SUMMARY:
Complications such as postoperative pain and delayed socket healing are relatively common following surgical extraction of mandibular third molars. Various biomaterials have been investigated to enhance wound healing and reduce postoperative morbidity. Hyaluronic acid (HA) has demonstrated anti-inflammatory and regenerative properties that may improve both soft and hard tissue healing.

The aim of this study is to evaluate the effect of topical hyaluronic acid on postoperative pain and alveolar socket bone healing following surgical extraction of mandibular third molars. A prospective, randomized, controlled clinical trial with a split-mouth design will be conducted. Twenty patients requiring bilateral mandibular third molar surgical extraction will be enrolled. In each patient, one extraction socket will receive hyaluronic acid combined with a collagen sponge, while the contralateral socket will receive a collagen sponge alone, according to random allocation. Postoperative pain will be assessed using a visual analogue scale, and socket healing will be evaluated radiographically and histologically.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, controlled clinical trial with a split-mouth design to assess the effect of topical hyaluronic acid on postoperative pain and alveolar socket bone healing following surgical extraction of mandibular third molars. The study will be conducted at the Oral and Maxillofacial Surgery and Preventive Dentistry clinics, Faculty of Dentistry, Jordan University of Science and Technology, Irbid, Jordan.

A total of 20 patients requiring bilateral surgical extraction of mandibular third molars will be enrolled. All participants will receive verbal and written information regarding the study procedures, and written informed consent will be obtained prior to participation. Randomization will be performed using a closed-envelope method. In each patient, one extraction site will be randomly allocated to receive hyaluronic acid gel combined with a collagen sponge (test site), while the contralateral site will receive a collagen sponge alone (control site).

The hyaluronic acid used in this study is a low-molecular weight sodium hyaluronate gel (Hyadent®, BioScience GmbH, Ransbach-Baumbach, Germany), supplied in sterile 1 mL syringes with blunt angulated cannulas. Each syringe contains sodium hyaluronate (14.0 mg), sodium chloride (6.9 mg), and water for injection. The formulation has modified viscosity and a short resorption time, allowing rapid absorption by the surrounding tissues.

All surgical procedures will be performed by a single experienced oral surgeon under standardized conditions. Preoperative evaluation includes medical and dental history, clinical examination, and panoramic radiography. Local anesthesia will be administered using an inferior alveolar nerve block with buccal infiltration of 2% lidocaine with 1:100,000 epinephrine. A standardized mucoperiosteal envelope flap will be raised for all procedures. Bone removal and tooth sectioning will be carried out when necessary using a low-speed handpiece under copious sterile saline irrigation.

After tooth removal, hyaluronic acid gel will be placed into the extraction socket at the test site and covered with a collagen sponge. Control sites will receive a collagen sponge alone. Primary closure will be achieved using 3-0 silk sutures. All patients will receive standardized postoperative instructions and medications. Sutures will be removed on postoperative day seven.

Postoperative pain will be assessed using a visual analogue scale (VAS) ranging from 1 (no pain) to 10 (worst pain imaginable). Participants will record pain scores at standardized time points: 12 hours after surgery (postoperative day 1), postoperative day 3, and postoperative day 7.

Radiographic assessment of socket healing will be performed using orthopantomogram (OPG) imaging in a randomly selected subgroup of participants approximately eight weeks after extraction. Radiographs will be obtained using standardized exposure parameters and processed under controlled conditions to ensure consistency.

Histological evaluation of socket healing will be conducted six weeks after extraction. Core biopsies will be obtained from both extraction sites under local anesthesia without flap reflection using a 3 mm diameter graded trephine bur. Harvested specimens will be fixed in formalin, decalcified, processed, and stained with hematoxylin and eosin. Digital images will be analyzed using image analysis software to calculate the percentage of woven bone within predefined regions of interest.

Statistical analysis will be performed using Statistical Package for the Social Sciences (SPSS) software. Descriptive statistics will be calculated for all variables. Comparative analyses will be conducted to evaluate differences in postoperative pain and woven bone formation between test and control sites, as well as changes in pain intensity over time.

ELIGIBILITY:
Inclusion Criteria:

Male and female participants aged 18 to 35 years

Presence of bilateral impacted mandibular third molars classified as Pell and Gregory Class II, Position B

Classified as American Society of Anesthesiologists (ASA) Physical Status I

Absence of active local infection at the surgical site (e.g., no swelling, trismus, hyperthermia)

Ability to maintain adequate oral hygiene

Ability to understand and provide written informed consent

Ability to read and understand Arabic or English

Willingness to comply with study procedures and follow-up visits

Exclusion Criteria:

History of systemic diseases such as diabetes mellitus, hypertension, gastric ulcer, or other significant medical conditions

Presence of severe or chronic illness requiring frequent hospitalization

Pregnant or breastfeeding individuals

History of cognitive or motor impairment that may interfere with study participation

Use of anti-inflammatory or analgesic medications within two weeks before surgery

Known allergy or hypersensitivity to nonsteroidal anti-inflammatory drugs (NSAIDs)

Current smoker

Use of anticoagulant therapy

Any condition that, in the investigator's judgment, may interfere with healing or study outcomes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | 12 hours (postoperative day 1), postoperative day 3, and postoperative day 7. Units of measure is VAS score (1-10).
  Postoperative pain intensity will be assessed using a visual analogue scale (VAS) ranging from 1 (no pain) to 10 (worst pain imaginable). Participants will record pain scores at standardized time points following mandibular third molar extraction.
Alveolar Socket Bone Healing | 6 weeks after tooth extraction. units of measure is percentage of woven bone area (%)
  Alveolar socket bone healing will be evaluated histologically by quantifying the percentage of woven bone formation within the extraction socket. Core biopsies will be obtained six weeks post-extraction and analyzed using digital histomorphometry. The percentage of woven bone area within predefined regions of interest will be calculated using ImageJ software.

OTHER OUTCOMES:
Radiographic Assessment of Socket Healing | Preoperative baseline and 6-8 weeks post-extraction
  Radiographic socket healing will be assessed descriptively using orthopantomogram (OPG) imaging. Standardized radiographs will be obtained preoperatively and approximately six to eight weeks post-extraction to evaluate changes in socket radiodensity.

CONTACTS AND LOCATIONS:
Overall Officials: Rola Habashneh, Professor, Study Chair — Jordan University of Science and Technology
Locations (1):
- Higher specialty training center, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
The data of the participants collected are clinical and we should take their consent for any future studies. As our IRB approval is limited to this study, we cant share these data.

REFERENCES:
- [Background] Domic D, Bertl K, Lang T, Pandis N, Ulm C, Stavropoulos A. Hyaluronic acid in tooth extraction: a systematic review and meta-analysis of preclinical and clinical trials. Clin Oral Investig. 2023 Dec;27(12):7209-7229. doi: 10.1007/s00784-023-05227-4. Epub 2023 Nov 15. PMID 37963982